CLINICAL TRIAL: NCT00477048
Title: Efficacy and Safety of a Saquinavir Based Regimen in HIV-1 Infected Thai Patients Who Have Chronic IDV Associated Nephrotoxicity.
Brief Title: Efficacy and Safety of SQV in Patients Who Have Chronic IDV Nephrotoxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Roche Pharma AG (Industry); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 027
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: IDV Associated Nephrotoxicity
Keywords: IDV nephrotoxicity
MeSH Terms: interventions — Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Replace Indinavir with SQV in patients with indinavir toxicity
  Interventions: Drug: Saquinavir

INTERVENTIONS:
Drug: Saquinavir — SQV/r 1000/100 BID + NNRTI or SQV/r 1600/100 OD + 2 NRTI

SUMMARY:
Efficacy and safety of a saquinavir (SQV) based regimen in HIV-1 infected Thai patients who have chronic indinavir (IDV) associated nephrotoxicity.

DETAILED DESCRIPTION:
Primary objective:

To determine whether a switch to a SQV can cause improvements in renal function in patients with chronic IDV associated nephrotoxicity without improvement after IDV dose reduction.

Secondary objective:

1. To describe the pathophysiology of chronic IDV associated renal impairment through renal biopsies at baseline and week 48
2. To describe the pathophysiology of chronic IDV associated renal impairment through renal tubular function at baseline and week 48
3. To determine whether a switch to an SQV can cause improvements in renal pathophysiology in patients with chronic IDV associated nephrotoxicity through renal biopsies performed at baseline and at weeks 48
4. To determine whether a switch to an SQV results in improvements in hypertension, lipid profiles and cutaneous side effects

ELIGIBILITY:
Inclusion Criteria:

* IDV containing regimen for more than 1 year and have creatinine more than 1.4 at least 6 months/abnormal renal imaging/abnormal urinary examinations
* Viral load less than 50 copies

Exclusion Criteria:

* Saquinavir intolerance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Viral load less than 50 copies/ml Improvement of renal functions and renal imaging | 48 weeks

SECONDARY OUTCOMES:
Metabolic and cutaneous profile | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org